CLINICAL TRIAL: NCT06833398
Title: Arthroscopic Simple Biceps Tenotomy Versus Anchor Tenotomy Technique, Clinical Outcome and Ultrasound Assessment
Brief Title: Comparison Between Arthroscopic Simple Biceps Tenotomy & Anchor Technique Tenotomy with Clinical and Ultrasound Assessment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Sayed Shehata, resident at the Orthopaedic and Trauma Surgery department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: biceps tenotomy technique
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-12

CONDITIONS: Simple Biceps Tenotomy; Anchor Tenotomy
Keywords: Arthroscopic biceps tenotomy; Long head of biceps tendon (LHB) Popeye deformity Ultrasound assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arthroscopic simple Biceps tenotomy (Experimental): This group undergoes a straightforward arthroscopic procedure to release the LHB tendon. The technique is quick and avoids the need for implants or prolonged rehabilitation. However, it carries a risk of cosmetic deformities, such as the "Popeye" sign, and potential biceps muscle cramps postoperatively.
- anchor tenotomy technique (Experimental): This group undergoes a novel anchor-based tenotomy technique. The procedure aims to prevent the Popeye deformity by anchoring the released tendon in a specific position. While technically more complex than simple tenotomy, it is designed to improve cosmetic outcomes and potentially reduce postoperative complications.
  Interventions: Procedure: Anchor Tenotomy Technique:

INTERVENTIONS:
Procedure: Arthroscopic Simple Biceps Tenotomy: — Arthroscopic Simple Biceps Tenotomy: This procedure involves an arthroscopic release of the LHB tendon from its attachment at the superior glenoid labrum. It is a quick and simple technique that does not require implants or extensive postoperative rehabilitation. The main drawback is the potential for developing a "Popeye" deformity, where the biceps muscle bulges due to distal migration, as well as occasional muscle cramps.
Procedure: Anchor Tenotomy Technique: — Anchor Tenotomy Technique: This is a novel arthroscopic method where, after releasing the LHB tendon, it is anchored in place to prevent distal migration. The goal of this technique is to avoid the Popeye deformity and improve cosmetic outcomes while maintaining functional integrity. This procedure is technically more challenging and may involve a longer operative time compared to simple tenotomy.
  Arms: anchor tenotomy technique

SUMMARY:
Comparison between arthroscopic simple biceps tenotomy & anchor tenotomy technique regarding clinical outcomes & ultrasound assessment

DETAILED DESCRIPTION:
This research compares two surgical techniques for addressing pathologies of the long head of the biceps (LHB) tendon: arthroscopic simple biceps tenotomy and anchor tenotomy. The LHB tendon, originating from the supraglenoid tubercle, plays a critical role in forearm supination, elbow flexion, and shoulder abduction. Pathologies affecting this tendon often cause significant shoulder pain, with surgical options including tenotomy and tenodesis. While simple tenotomy is quick and avoids implant complications, it may result in cosmetic deformities like the "Popeye" sign and muscle cramps. Anchor tenotomy, a novel technique, aims to minimize these issues by preventing the Popeye deformity. This study employs a prospective randomized double-blinded controlled trial design at Assiut University Hospitals, involving 72 patients with LHB pathologies such as tendinitis, rotator cuff tears, and subacromial impingement. Exclusion criteria include prior tenodesis or neuromuscular diseases. Clinical outcomes will be assessed using functional scores (e.g., Oxford Shoulder Score), ultrasound evaluation of tendon positioning, and follow-up examinations at intervals up to one year post-surgery. The primary outcome focuses on the presence of the Popeye deformity, while secondary outcomes include postoperative shoulder function and tendon distalization measured via ultrasound. This research aims to provide evidence-based insights into the comparative effectiveness of these two techniques in improving clinical outcomes and minimizing complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with LHB pathologies such as :

Biceps tendinitis Rotator cuff tears Subacromial impengiment Instability & traumatic causes

Exclusion Criteria:

* LHB Tenodesis Patients with neuromuscular disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
evaluate for popeye sign after arthroscopic simple biceps tenotomy vs anchor technique tenotomy | 1 year
  clinical evaluation of shoulder function postoperative by dynamometer & US assessment of LHB tendon distalization after LHB tenotomy .
  Remove

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No